CLINICAL TRIAL: NCT07101575
Title: Cardiac Observational Study of Patients With Hereditary Hemorrhagic Telangiectasia
Brief Title: Cardiac Evaluation in Hereditary Hemorrhagic Telangiectasia
Acronym: CARDI-HHT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7459
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Transthoracic echocardiography with bubble test, by intravenous infusion of agitate saline solution

SUMMARY:
Hereditary haemorrhagic telangiectasia (HHT) is a rare autosomal dominant genetic disease associated with mutations in genes encoding proteins of the transforming growth factor β (TGF-β) family, i.e. endoglin (ENG), activin receptor A (ACVRL1), and SMAD 4 (small mother against decapentaplegic 4). Mutations in any of these genes lead to the onset of arteriovenous malformations (AVMs). The clinical consequences of this syndrome are primarily AVM-associated complications.

Major cardiovascular consequences occur in the more advanced stages, but their prevalence is low. Most HHT patients are asymptomatic, and ischemic heart disease has a significantly lower prevalence than in the general population. The limited sample size of studies currently published in the literature makes it difficult to characterize any subclinical cardiovascular alterations in asymptomatic HHT subjects.

Alterations in TGF-β family proteins likely result in a protective effect on the coronary circulation against atherosclerosis. A thorough understanding of the potential protective factors against coronary artery disease, underlying HHT alterations, may allow the development of gene therapy models inspired by the HHT phenotype. Some manifestations of extracellular matrix remodelling at the tissue level (i.e. myocardial and valvular) may be more prevalent in HHT patients than in the general population. Finally, any subclinical alterations in cardiac function related to chronic anaemia and possible iron overload due to iron replacement therapy are not yet known.

Primary objective of the study will be to perform a complete echocardiographic characterization, using new imaging methods aimed at identifying even subclinical dysfunctions of cardiac mechanics, including a phenotyping of the morphology and function of the valvular systems, as well as paradoxical shunts.

Secondary objectives of the study will be: 1) To verify whether there are echocardiographic differences, related to extracellular matrix remodelling, in addition to the presence of shunts, between the various HHT genotypes and to identify any genotype-phenotype correlations. 2)To verify the impact of chronic anaemia and iron supplementation on cardiac mechanics in relation to possible genotype-phenotype interactions.

About study methodology, collection and analysis of clinical and echocardiographic data will be obtained from routine cardiac assessments performed as part of the HHT clinical-care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 10 years of age with a genetic diagnosis, i.e. a pathogenic mutation in the endoglin (ENG), activin receptor A (ACVRL1) or small mother against decapentaplegic (SMAD4) gene, and/or a clinically confirmed diagnosis of hereditary hemorrhagic teleangectasia (HHT) according to the Curaçao criteria
* Signed informed consent

Exclusion Criteria:

* Patients whose echocardiographic images are of suboptimal quality and cannot be adequately analysed.
* No signed informed consent

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 380 patients will be enrolled, approximately 30 of whom are between the ages of 10 and 18. These patients currently undergo echocardiography with bubble test for pulmonary arteriovenous malformation (AVM) screening, as part of the hereditary haemorrhagic telangiectasia (HHT) clinical care pathway and therefore as part of standard clinical practice. Pregnant women and paediatric patients (aged 10 and older) will constitute subgroups and will be analysed separately.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2030-08-05 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of suclinical cardiac mechanical dysfunction | 30 minutes
  Perform a comprehensive echocardiographic characterization, using new imaging techniques to identify even subclinical cardiac mechanical dysfunction, including phenotyping of the morphology and function of the valvular systems, as well as paradoxical shunts

SECONDARY OUTCOMES:
Genotype-phenotype correlations | 6 months
  Verify whether there are echocardiographic differences related to extracellular matrix remodelling, in addition to the presence of shunts, between the various hereditary hemorrhagic telangiectasia (HHT) genotypes and identify any genotype-phenotype correlations
Impact of chronic anaemia | 6 months
  Verify the impact of chronic anaemia and iron supplementation on cardiac mechanics in relation to possible genotype-phenotype interactions

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Locorotondo, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS Roma